CLINICAL TRIAL: NCT04320407
Title: A Post-market Interventional Cohort Study Evaluating the Clinical Efficacy of the Osia 2 System in the US Market.
Brief Title: Osia CPT Code Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5778
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-09

CONDITIONS: Conductive Hearing Loss; Mixed Hearing Loss
Keywords: conductive hearing loss; mixed hearing loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Osia 2 System (Experimental): Osia 2 Active Osseointegrated Implant System for Bone Conduction
  Interventions: Device: Osia 2 System

INTERVENTIONS:
Device: Osia 2 System — The external Sound Processor, Osia 2 Active Osseointegrated Implant System for Bone Conduction, captures and digitizes the sound which is transferred to the internal implant where it is converted to an electrical signal.

SUMMARY:
To evaluate the clinical efficacy of the Osia 2 system in patients with conductive or mixed conductive hearing loss in a US cohort.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Proficient in English.
* Hearing loss etiology of Conductive or Mixed Conductive loss.
* Bone conduction PTA (.5, 1, 2, and 3 kHz) better than or equal to 55 dB HL in the treatment ear.
* Aged 18 years and older.

Exclusion Criteria:

* Unwilling to wear the treatment device or comply with the surgical and rehabilitation requirements of the study.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Medical, audiological or psychological conditions, as judged by the investigator that might contraindicate participation in the clinical investigation.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or contractors engaged by Cochlear for the purposes of this investigation.
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.
* Prior experience with a surgical bone conduction treatment option
* Insufficient bone quality to support the BI300 implant as determined by the surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Syms, MD, Principal Investigator — Arizona Hearing Center
Locations (4):
- United States (4):
  - Arizona Ear Center, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - University of Michigan, Ann Arbor, Michigan
  - Center for Hearing and Balance, Chesterfield, Missouri

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Osia 2 System
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Osia 2 System
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adaptive Speech in Noise Test Score for Osia 2 System at 3 Months Post-surgery
Description: Assessed with the Quick SIN test preoperative and at 3 months post-surgery. The Quick SIN test has a score range from +25.5 dB (decibel) SNR (signal-to-noise ratio) to -5 dB SNR. The participants are tested on 4 tests lists; each consists of 6 sentences (with 5 key words per sentence) that are presented at signal-to-noise ratios (SNR) which are decreased manually in 5-dB steps from 25 to 0. The key words in sentences are scored and counted as correct from an easy to difficult or unfavorable SNR. The best possible score on this test would be that of -5 dB SNR where all of the key words are repeated back correctly as a function of the SNR. The mean unaided preoperative score is substracted from the aided score at 3 months. A lower score indicates a better performance.
Time Frame: Preoperative, 3 months post-surgery
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Osia 2 System
Number analyzed (Participants) | 20
Score on a scale | 6.1 (6.9)

2. Secondary Outcome: Number of Device or Procedure Related Adverse Events
Description: A device or procedure related adverse event (AE) is an AE for which a causal relationship between the use of the medical device and the AE cannot be ruled out. All related AEs are reported.
Time Frame: 6 months post-surgery
Measure: Number; unit: Number of events
Arm/Group | Osia 2 System
Number analyzed (Participants) | 20
Number of events | 15

ADVERSE EVENTS:
Time Frame: From the day of surgery (day 0) to 6 months post-surgery
Description: Adverse events with a frequency threshold > 5% are reported.
Arm/Group | Osia 2 System
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Osia 2 System (N=20)
Post-operative pain (General disorders) | 5 (5)
Post-operative swelling (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can't publish or discuss the results without the permission of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04320407/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT04320407/SAP_001.pdf